CLINICAL TRIAL: NCT03944044
Title: Paracetamol Route in Palliative Care Patients : Intravenous Versus Subcutaneous Route Pharmacokinetics, Study Protocol for a Randomized Equivalence Pilot Trial
Brief Title: Paracetamol Route in Palliative Care Patients (PARASCIVPALLIA)
Acronym: PARASCIVPALL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17-245
Record Dates: First submitted 2019-01-25; First posted 2019-05-09 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Palliative Care
Keywords: Paracetamol; Acetaminophen; Palliative care; Subcutaneous administration; intravenous administration; pharmacokinetic

STUDY DESIGN:
Intervention Model Description: This is a comparative, randomized, open, crossover, bicenter clinical trial with SC and IV paracetamol injections successively given to each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous route first (Other): The first route of administration is designated by randomization. In the subcutaneous group, patients received intravenous route in a second time.
  Interventions: Other: Paracetamol route in palliative-care patients: intravenous versus subcutaneous route Pharmacokinetics study protocol
- Intravenous route first (Other): The first route of administration is designated by randomization. In the intravenous group, patients received subcutaneous route in a second time.
  Interventions: Other: Paracetamol route in palliative-care patients: intravenous versus subcutaneous route Pharmacokinetics study protocol

INTERVENTIONS:
Other: Paracetamol route in palliative-care patients: intravenous versus subcutaneous route Pharmacokinetics study protocol — Compare the pharmacokinetic (PK) of SC and intravenous (IV) routes in the same patient in a palliative care situation, to determine if there is a PK equivalence between these two modes of administration of Paracetamol.

SUMMARY:
Background: Among palliative-care patients, subcutaneous route is often an alternative to intravenous route yet pharmacological and clinical data are lacking. Many French palliative crew are now using empirically paracetamol by subcutaneous route also there is no data to support this practice. The aim of the present study is to compare pharmacokinetics parameters between intravenous and subcutaneous route for palliative-care patients.

Methods/design: A randomized, open, crossover, bicenter study in two palliative care centers. The aim is to demonstrate the pharmacokinetic equivalence between the two routes of administration. Data analysis will be performed by Wilcoxn's signed Rank Test with an alpha risk of 5 percent. All adverse events will be reported for a safety analysis.

Discussion: This trial may permit, if a pharmacokinetic equivalence is established, to build randomized controlled trials to then assess the efficacy and tolerability of subcutaneous paracetamol administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old, hospitalized
* Patients in a palliative care situation
* Patients having an intravenous device with the presence of a venous reflux (be implantable venous site, picc-line, central track)
* Patients having a spontaneous pain, not related to care, with a numeric pain rate scale (NPRS) > 3/10 or have a systematic prescription of paracetamol in the usual treatment
* Patients able to do an auto-evaluation of their pain by NPRS
* No contraindications of paracetamol
* No contraindications of alternative antalgic (low opioids, strong opioids, Non-steroidal anti-inflammatory)
* Possibility to not take paracetamol in the previous 24 hours before inclusion
* Patients with a blood test dating back less than 7 days, with no severe renal or hepatic failure
* Patients related with a French social security regime
* Patients accept to participate in the study, with written consent.

Exclusion Criteria:

* Patients under legal protection
* Patients who participate in another study less than 30 days before
* Patients weighing less than 50 kg
* Patients having a contraindication to subcutaneous route
* Pregnant or breastfeeding woman
* Patients who having a paracetamol administration less than 24 hours before the beginning of the inclusion
* Patients who having a low opioid less than 2 hours before or a strong opioid less than one hour before the beginning of administration of paracetamol
* Patients having a fever
* No possibility of communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
paracetamolemia dosage after intravenous route | At injection time
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 15 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 60 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 90 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 120 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 240 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 360 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after intravenous route | 480 minutes after injection
  measurement of paracetamol blood concentration after intravenous route
paracetamolemia dosage after subcutaneous route | at injection time
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 15 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 30 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 45 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 60 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 90 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 120 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 240 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 360 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route
paracetamolemia dosage after subcutaneous route | 480 minutes after injection
  measurement of paracetamol blood concentration after subcutaneous route

SECONDARY OUTCOMES:
pain scale | at injection time
  numeric sale (0-10)
pain scale | 15 minutes after injection time
  numeric sale (0-10)
pain scale | 60 minutes after injection time
  numeric sale (0-10)
pain scale | 90 minutes after injection time
  numeric sale (0-10)
pain scale | 120 minutes after injection time
  numeric sale (0-10)
pain scale | 240 minutes after injection time
  numeric sale (0-10)
pain scale | 360 minutes after injection time
  numeric sale (0-10)
pain scale | 480 minutes after injection time
  numeric sale (0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Caen, France

REFERENCES:
- [Derived] Vernant M, Lepoupet M, Creveuil C, Alix A, Gourio C, Peyro-Saint-Paul L, Lelong-Boulouard V, Guillaume C. Intravenous versus subcutaneous route pharmacokinetics of paracetamol (acetaminophen) in palliative care patients: study protocol for a randomized trial (ParaSCIVPallia). Trials. 2020 Feb 4;21(1):138. doi: 10.1186/s13063-019-3969-0. PMID 32019598